CLINICAL TRIAL: NCT01303731
Title: Phase IV, Randomized, Parallel Designed, Single Blinded Study, Comparing the Standard and Minidose Spinal Anesthesia Using Marcaine Spinal 0.5% Heavy With Addition of Fentanyl During Cesarean Section
Brief Title: Comparison of Standard and Minidose Spinal Anesthesia for Cesarean Section Operation Using Marcaine Spinal 0.5% Heavy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Dr Boris Yanovsky, Bnai Zion Medical Center, Haifa, Israel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0123-10-BZ
Record Dates: First submitted 2011-01-20; First posted 2011-02-25 (Estimated); Last update posted 2011-02-25 (Estimated); Status verified 2011-01

CONDITIONS: Cesarean Section; Anesthesia, Spinal; Local Anaesthetics Causing Adverse Effects in Therapeutic Use
Keywords: Spinal anesthesia; Cesarean section; Marcaine Spinal 0.5% Heavy minidose; Fentanyl; Local Anesthetics
MeSH Terms: interventions — Bupivacaine; Fentanyl

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Standard dose Marcaine Spinal 0.5% Heavy (Active Comparator): Standard group - will receive spinal anesthesia induced by Marcaine Spinal 0.5% Heavy 12.5 mg (2.5 ml).
  Interventions: Drug: Bupivacaine
- Minidose of Marcaine Spinal 0.5% Heavy (Experimental): Minidose group - will receive spinal anesthesia induced by Marcaine Spinal 0.5% Heavy 7.5 mg (1.5 ml) diluted in 0.75ml of patient's CSF (0.25 ml)with addition of Fentanyl 12.5 mcg (total 2.5 ml)
  Interventions: Drug: Bupivacaine and Fentanyl

INTERVENTIONS:
Drug: Bupivacaine and Fentanyl — Spinal anesthesia with Marcaine Spinal 0.5% Heavy 7.5 mg (1.5 ml) diluted in 0.75ml of patient's CSF (0.25 ml)with addition of Fentanyl 12.5 mcg (total 2.5 ml)
  Other Names: Marcaine Spinal 0.5% Heavy; Fentanyl-Janssen
  Arms: Minidose of Marcaine Spinal 0.5% Heavy
Drug: Bupivacaine — Spinal anesthesia with Marcaine Spinal 0.5% Heavy 12.5 mg (2.5 ml)
  Other Names: Marcaine Spinal 0.5% Heavy
  Arms: Standard dose Marcaine Spinal 0.5% Heavy

SUMMARY:
The objectives of this study is to test a combination of low dose local anesthetic Bupivacaine diluted in patient's CSF with lipophilic opiate Fentanyl for optimal spinal anesthesia during Cesarean Section. The dilution of Bupivacaine with CSF in our study would result in effective spinal anesthesia with relatively limited motor block, quick recovery of motor function and relatively long lasting analgesia. We expect lower incidence of side effects with this combination than with convenient dose of Bupivacaine.

DETAILED DESCRIPTION:
Spinal anesthesia is the most frequent type of anesthesia used for Cesarian Section. However, despite decades of safe utilization there is still controversy about the best combination of local anesthetics and additives needed to obtain the optimal result. The objectives of this study is to test a combination of low dose local anesthetic Bupivacaine diluted in patient's CSF with lipophilic opiate Fentanyl for compliance with the criteria of optimal spinal anesthesia. Bupivacaine is the most frequently used local anesthetic in the last twenty years . It characterized by fast onset, high potency and long action . Albeit this is intrinsic characteristic of specific local anesthetic, its manifestation can be affected by concentration. It has been shown that dilution of local anesthetic with CSF can result in sensory block with less profound motor block.

Thus dilution of Bupivacaine with CSF in our study would serve double function: it would speed the recovery from the spinal anesthesia and minimize the expression of the motor block.Addition of opiates to local anesthetics has been widely used . It has been shown that this addition improves quality of spinal anesthesia and prolongs analgesia without significant prolongation of recovery from motor block.

In summary, we would use well known safe local anesthetic Bupivacaine in low dose and low concentration (after dilution with patient's CSF) in conjunction with highly lipophilic opiate Fentanyl. We suppose it will result in effective spinal anesthesia with relatively limited motor block, quick recovery of motor function and relatively long lasting analgesia. We expect lower incidence of side effect with this combination than with convenient dose of Bupivacaine.

Good pain relief and swift restoration of ability to ambulate will be important for prevention of postoperative complications, will diminish the need for systemic analgetic drugs that can affect nursing and will increase patients' satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Women over 38 weeks of pregnancy, who read and write Hebrew
* ASA class I and II
* Age between 18 and 40 years
* Weight 50-100 kg
* Elective Cesarean Section for singlet pregnancy

Exclusion Criteria:

* Previous history of two or more Cesarean Sections
* Contraindications for regional anesthesia
* Active pain before surgery
* Non singlet pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
prominence of motor blockade | up to 2 h
  At the begining of the surgery and at the entry of the patients to PACU motor block will be evaluated

SECONDARY OUTCOMES:
operative condition | up to 1 h
  Upon completion of surgery attending surgeon will be asked to rate the operative condition.
intraoperative hypotension | up to 1 h
  Number of treatments for hypotensions during the surgery will be monitored.
need for postoperative pain medication | up to 2 h
  The pain or discomfort intensity during the surgery, and at PACU will be graded.
general patient satisfaction | after 24 h
  On the next day, all patients will be asked to rate their satisfaction following the anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Boris Yanovsky, MD, Principal Investigator — Bnai Zion Medical Center, Haifa, Israel
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel